CLINICAL TRIAL: NCT07057661
Title: Evaluation of Difficult Airway in Adenotonsillectomy Patients With Ultrasound
Brief Title: Evaluation of Difficult Airway With Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Tuba Kuvvet Yoldaş, MD, Anesthesia Specialist, Izmir City Hospital
Other Study IDs: İSH-ANS-TK-02
Record Dates: First submitted 2025-06-08; First posted 2025-07-10 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Adenotonsillectomy Surgery
Keywords: airway management; pediatric patients; ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Pediatric patients who underwent adenotonsillectomy
- Group 2: Pediatric patients who underwent any surgical operation

SUMMARY:
An unexpected difficult airway can lead to severe hypoxia and even death. Accurate airway assessment can reduce the incidence of difficult endotracheal intubation and related complications. Studies have shown that some ultrasonic indicators can predict difficult airways in adults to some extent. Studies have begun to investigate whether ultrasonic parameters can be used to predict difficult airways in children.Ultrasonic measurements of certain airway parameters have predictive value for difficult airways; therefore, airway ultrasonography is recommended as an aid in difficult airway prediction. We think that in pediatric patients with adenotonsillectomy, we will encounter more difficult airway because there may be anatomical differentiation due to adenoid and tonsillar hypertrophy. We aimed to evaluate the frequency of difficult airway with USG measurements in pediatric patients undergoing adenotonsillectomy.

Group 1:Pediatric patients who underwent adenotonsillectomy Group 2: Pediatric patients who underwent any surgical operation We will evaluate two patient groups.

DETAILED DESCRIPTION:
Ultrasonography (USG) is widely used in airway management, such as prediction of difficult airways, localization of cricothyroid membranes, selection of tracheal tubes, and evaluation of patients with a full stomach. Among these, ultrasonic measurements of the dimensions of certain airway parameters have predictive value for difficult airways; therefore, airway ultrasonography is recommended as an aid in difficult airway prediction. Many studies have shown that some ultrasonic parameters such as hyomental distance in the extension position and distance from the skin to the epiglottis can predict difficult airways in adults. However, it is unclear whether these parameters can be used to predict difficult airways in children. In recent studies, various protocols have started to be established . We think that we will encounter more difficult airways in pediatric patients with adenotonsillectomy because there may be anatomical differentiation due to adenoid and tonsillar hypertrophy. Therefore, we will evaluate the relationship between skin-epiglottic distance, hyomental distance and tongue base thickness measurements, which are used in most studies, and the mallampati score on physical examination and the Cormack Lehane score during laryngoscopy. The aim of this study was to compare the frequency of difficult airway between pediatric patients who underwent adenotonsillectomy (Group 1) and pediatric patients who underwent any surgical operation (Group 2) using USG measurements.

Group 1:Pediatric patients who underwent adenotonsillectomy Group 2: Pediatric patients who underwent any surgical operation

ELIGIBILITY:
Inclusion Criteria:

1. ASA 1-2 patients
2. Pediatric patients aged 3-8
3. Those planned for elective surgery

Exclusion Criteria:

1. Those with a history of congenital anomalies (head, face, body)
2. ASA 3-4-5 patients
3. Those who will undergo emergency surgery
4. Those who will be subjected to an airway or anesthesia technique other than orotracheal intubation
5. Newborn group patients
6. Patients younger than 3 years old and older than 8 years old

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who underwent adenotonsillectomy and any surgical operation
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
DSE: Distance from skin to epiglottis | Preoperative , before the administration of anesthesia
  the vertical distances from the submental skin to the midpoint of the epiglottis
HMDE: Hyomental distance in the extended position | Preoperative , before the administration of anesthesia
  the distance from the lower border of the mentum of the mandible to the upper border of the hyoid bone
Tongue base thickness | Preoperative , before the administration of anesthesia

SECONDARY OUTCOMES:
Cormark Lehane score | During laryngoscopy
  Grade 1: being a full view of the glottis Grade 2 : being a partial view Grade 3: being only a view of the epiglottis Grade 4: being an absent view of the glottis and epiglottis

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Kuvvet Yoldas, MD, Anesthesiology Specialist, Principal Investigator — Izmir City Hospital
Locations (1):
- İzmir City Hospital, Izmir, Bayraklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No